CLINICAL TRIAL: NCT05909930
Title: Effectiveness of TheRApeutic ExercIse aNd EDucation on Patients With Massive Rotator Cuff Tears (the TRAINED Study): a Multicenter Non-controlled Trial
Brief Title: Effectiveness of TheRApeutic ExercIse aNd EDucation on Patients With Massive Rotator Cuff Tears
Acronym: TRAINED
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial support for the project has been discontinued.
Sponsor: Hospital Universitario Fundación Alcorcón (Other)
Collaborators: Hospital Universitario La Paz (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario La Princesa (Unknown); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Principe de Asturias (Other); Hospital Universitario de Fuenlabrada (Other); Hospital Universitario Infanta Leonor - Vallecas/H. Virgen de la Torre (Unknown)
Responsible Party: Principal Investigator, Rubén Fernández Matías, Principal Investigator, Hospital Universitario Fundación Alcorcón
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23/68
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Injuries
Keywords: Physical therapy; Massive rotator cuff tear; Therapeutic resistance exercise; Multicenter
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic exercise and education (Experimental): The treatment will consist of a progressive resistance exercise program along with education.
  Interventions: Other: Therapeutic resistance exercise; Other: Education

INTERVENTIONS:
Other: Therapeutic resistance exercise — Therapeutic exercise program based on individualized progressive resistance exercises performed during 6 months at home, with a frequency of 1-3 sessions per week at the hospital.
Other: Education — Education applied during all the therapeutic process, focusing on diverting the patient's attention away from the structural lesion, explaining the relationship between pain/disability and tissue injury, explaining the meaning of pain during exercises, and explaining the objectives of the implemented treatments.

SUMMARY:
The aim of this multicenter non-controlled study will be to evaluate the effectiveness of a physical therapy treatment based on resistance exercise and education for patients with massive rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

* Massive rotator cuff tear diagnosed by ultrasound imaging or magnetic resonance imaging. The definition of massive will be the rears including 2 or more tneonds, or the ones with an extension equal or greater to 5cm in the short or long axis.
* To have a degree of disability equal or greater to 15% in the Oxford Shoulder Score.
* Adequate comprehension of written and spoken Spanish

Exclusion Criteria:

* Loss of passive external rotation at 0º of shoulder abduction equal or greater to 50% compared to contralateral side.
* Suspected neck-related shoulder pain.
* Suspected visceral-related shoulder pain.
* Humerus and/or scapular fractures within the last year.
* Previous rotator cuff repair surgery within the last year.
* Presence of cancer, fibromyalgia, neurological and/or other systemic diseases.
* Cognitive impairment that makes it impossible to perform therapeutic exercise.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Shoulder disability | Baseline, change from baseline to 3-month, change from baseline to 6-month, and change from baseline to 1-year.
  Shoulder disability measured with the Oxford Shoulder Score, which ranges from 0 (no disability) to 100 (maximum degree of disability).

SECONDARY OUTCOMES:
Shoulder pain intensity | Baseline, change from baseline to 3-month, change from baseline to 6-month, and change from baseline to 1-year.
  Shoulder pain intensity measured with a numeric pain rating scale, which ranges from 0 (no pain) to 10 (worst imaginable pain).
Need for surgery | 3-month, 6-month, and 1-year.
  Need for surgery for the rotator cuff tear registered as a dichotomous variable (YES/NO).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
IPD data will be shared with other researchers upon reasonable request.